CLINICAL TRIAL: NCT00656279
Title: Intensive Patient Education Using the Phosphorus Point System© Tool to Improve Serum Phosphorus Levels in Patients With Chronic Kidney Disease
Brief Title: Intensive Dietary Education to Lower Serum Phosphorus in Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMH07-377
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; predialysis; hyperphosphatemia; dietary intervention; intensive dietary education; low phosphorus diet
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intensive dietary phosphorus education
  Interventions: Behavioral: Intensive dietary phosphorus education
- 2 (No Intervention): Standard dietary education consists of the dietitian assessing laboratory values and dietary intake and providing dietary education for abnormal values using handouts developed for specific nutrients.

INTERVENTIONS:
Behavioral: Intensive dietary phosphorus education — Intensive dietary phosphorus education will be completed using the Phosphorus Point System Tool, a booklet listing phosphorus points for food items based on the phosphorus content. Patients will be allotted a maximum of 32-40 phosphorus points daily. Points consumed will be tracked by the patients via daily tracking sheets which require patients to list the phosphorus food items consumed, the number of points, and the time and amount of phosphate binders. Patients in this group will also receive intensive education about phosphorus additives. As a part of the program that supports the tool, patients will receive weekly telephone calls for the first 6 weeks to address any questions about the tool and find phosphorus point values of foods not listed within the tool.
  Arms: 1

SUMMARY:
A low phosphorus diet is recommended for patients with chronic kidney disease who exhibit high levels of phosphorus. The purpose of this study is to determine the effects of a more intensive, innovative dietary phosphorus educational intervention on reducing serum phosphorus levels, as well as improving dietary adherence, dietary satisfaction and phosphorus knowledge level in patients with chronic kidney disease.

DETAILED DESCRIPTION:
High serum phosphorus concentration (hPhos) commonly occurs in chronic kidney disease (CKD) secondary to declining renal function. hPhos increases the risk of developing metastatic calcification, secondary hyperparathyroidism, renal osteodystrophy and cardiovascular complications. Patients with hPhos are advised to restrict their dietary phosphorus intake to 800-1000mg/d, as per National Kidney Foundations'Kidney Disease Quality Outcomes Initiative (KDOQI). Adherence to a phosphorus restricted diet is often challenging for CKD patients, as they may be required to follow various dietary restrictions, and there is significant quantities of hidden phosphorus in processed foods. This randomized controlled trial is designed to compare the effectiveness of more intensive phosphorus education (IPE) using the innovative Phosphorus Point System Tool© versus standard phosphorus education (SPE) using the Choose/Avoid list on 1) serum phosphorus levels (primary outcome) 2) dietary adherence, dietary knowledge and satisfaction in patients with pre-dialysis CKD. We hypothesize that patients receiving IPE will have lower serum phosphorus than those receiving SPE. Fifty patients attending a pre-dialysis CKD clinic with serum phosphorus > 1.49 mmol/L will be randomly assigned to IPE or SPE and followed over 12 weeks. Serum phosphorus, dietary intakes using the 5-pass repeat 24-hour dietary recall method, dietary knowledge and satisfaction by validated questionnaires, will be measured at baseline, 6 weeks and 12 weeks. The study's findings on the impact of more intensive innovative dietary phosphorus education in patients with pre-dialysis CKD will serve towards developing best practice of care and potentially reduce long-term complications.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Patient with pre-dialysis CKD attending the Progressive Renal Disease Clinic (PRDC) at St. Michael's Hospital
* Six-month mean serum phosphorus > 1.35 mmol/L
* Able to provide informed consent

Exclusion Criteria:

* Currently on dialysis
* Current malignancy
* Inability to use Phosphorus Point System (PPS) Tool

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Serum phosphorus | baseline, week 6, week 12

SECONDARY OUTCOMES:
Dietary adherence | baseline, week 6, week 12
Dietary satisfaction | baseline, week 6, week 12
Phosphorus management knowledge-level | baseline, week 6, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Darling, PhD, Principal Investigator — St. Michael's Hospital & University of Toronto
Locations (1):
- St. Michael's Hospital Progressive Renal Disease Clinic, Toronto, Ontario, Canada